CLINICAL TRIAL: NCT04426747
Title: Impact of Barriers and Facilitators to Physical Activity in Patients With Inflammatory Arthritis and Link With Physical Activity Collected by Mobile Phone Apps: a Cross-sectional Study
Brief Title: Impact of Barriers and Facilitators to Physical Activity in Patients With Inflammatory Arthritis
Acronym: ImBAIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Laure Gossec, Clinical Professor, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: 2019
Record Dates: First submitted 2019-12-05; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Inflammatory Arthritis; Ankylosing Spondylitis; Rheumatoid Arthritis; Psoriatic Arthritis
Keywords: Physical activity; Barriers; Facilitators
MeSH Terms: conditions — Arthritis; Spondylitis, Ankylosing; Arthritis, Rheumatoid; Arthritis, Psoriatic; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Background: Patients with inflammatory arthritis (IA), such as spondyloarthritis (axSpA), rheumatoid arthritis (RA) or psoriatic arthritis (PsA) are more prone to physical inactivity but derive specific benefits from regular physical activity. Barriers and facilitators to physical activity (B&F-PA) are key elements and knowledge of their correlation to physical activity is essential for developing interventions to promote physical activity that have a greater likelihood of success.

Objectives: primary objective will be to measure the correlation of these B&F-PA to physical activity collected through apps. Secondary objective will be to (I) to quantify physical activity collected through apps in IA patients and (II) to observe the link between physical activity, B&F to physical activity and adherence to treatment.

Patients and methods: This is an international, multicentric, cross-sectional study.

Patients: From the first of September to the first of February 2020, all patients with definite axSpA, RA or PsA, aged above 18 and able to walk, who have a mobile phone compatible with apps that can track steps, who agree to participate and give his oral informed consent and with ability to read and write in the language of the participating country, seen in outpatient visits in the participating centers, will be asked to participate. The planed inclusion was 200 participants.

Data collection: clinical data and information about physical activity and B&F-PA will be entered by rheumatologists during or electronically by patients at the same time point.

Questionnaire for B&F-PA: a patient reported questionnaire was recently developed for this study in 2019 based on a systematic review to identify the main B&F-PA. A list of questions was generated from the systematic review reviewed and tested for face validity by 11 experts and confronted to 20 patients with IA through a cognitive debriefing.

Physical activity: Physical activity will be measured objectively during the last 7 days by apps already installed by default on the mobile phone of participants and subjectively with the International Physical Activity Questionnaire short version (IPAQ-S).

Other outcomes: Stage of exercise behavior change and adherence to treatment will also be collected.

Planned analyses: Perceived B&F-PA will be described using frequencies. A score will be calculated for each participant representing the limitations or facilities to perform physical activity.

Analysis of the physical activity: The distribution of mean number of steps will be assessed visually for outliers. Univariate analysis will be completed between mean number of steps and gender, age, disease and stages of change. Correlation between mean number of steps and IPAQ-S score will be calculated.

Link between physical activity and barriers and facilitators: The link between B&F questionnaire score and mean number of steps will be tested using linear regression. Then multivariate regression including demographic variables, psychological status and disease characteristics will be performed.

Outcomes of the study: The expected outcomes of the ImBAIA study are a better understanding of B&F to physical activity in patients with IA and their impact to limit or to favor physical activity. We also expect to observe the level of physical activity of an IA population objectively measured with apps. Finally, a validation was expected to use questionnaire of B&F.

ELIGIBILITY:
Inclusion Criteria:

* aged above 18 and able to walk
* Definite IA confirmed by the rheumatologist and based on usual criteria: axSpA (referring to the Assessment of Spondyloarthritis international Society classification criteria (51)), RA (referring to the international classification criteria of RA (52)) or PsA (referring to the ClASsification of Psoriatic Arthritis (CASPAR) criteria (53)), with no restriction for co-morbidities,
* have a mobile phone compatible with apps that can track steps,
* agree to participate and give informed consent,
* ability to read and write in the language of participating country.

Exclusion Criteria:

Patients who don't speak or read the local language or are not comfortable filling in a Case Report Form in the local language or who don't have a mobile phone compatible with health apps.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Outpatients from secondary and tertiary care hospitals in France and in the United Kingdom will be invited to participate. Over the 5 months recruitment period, all patients with definite axSpA, RA or PsA who satisfy the inclusion criteria, seen in outpatient visits in the participating centers by one of the investigators, will be asked to participate. We plan to include 200 participants (based on a sample size calculation explained in statistical analysis part), 10-20 patients in each center, with a maximum of 30 patients per center and a competitive recruitment. We will aim for a minimum of 50 patients per disease group. After including of 50% of the population we will reorient inclusion if needed. Data will be collected at a single moment, during a usual visit.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-11-16 (Actual); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Physical activity (mean steps per day on the last full week (1 week) at inclusion) | Collected on the last full week at inclusion
  Physical activity objectively measured by patient's mobile phone at inclusion during the last full week (1 week)

CONTACTS AND LOCATIONS:
Locations (1):
- Laure Gossec, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davergne T, Tekaya R, Sellam J, Tournadre A, Mitrovic S, Ruyssen-Witrand A, Hudry C, Dadoun S, Avouac J, Fautrel B, Gossec L. Influence of perceived barriers and facilitators for physical activity on physical activity levels in patients with rheumatoid arthritis or spondyloarthritis: a cross-sectional study of 150 patients. BMC Musculoskelet Disord. 2021 Oct 30;22(1):915. doi: 10.1186/s12891-021-04792-7. PMID 34717606